CLINICAL TRIAL: NCT03234517
Title: Continuous Versus Interrupted Use.of Vaginal Probiotic Plus Vaginal Clindamycin Cream for Bacterial Vaginosis a Randomized Controlled Study
Brief Title: Vaginal Clindamycin Cream Plus Vaginal Probiotic for Bacterial Vaginosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, IBRAHIM ABD ELGAFOR, assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zuh- 8
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2017-07

CONDITIONS: Bacterial Vaginosis Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal Clindamycin Cream Plus continuous Vaginal Probiotic (Experimental): Vaginal Clindamycin Cream followed by continuous Vaginal Probiotic use for 60 days
  Interventions: Drug: Vaginal Clindamycin Cream; Drug: Vaginal Probiotic
- Vaginal Clindamycin Cream Plus interrupted Vaginal Probiotic (Active Comparator): Vaginal Clindamycin Cream followed by interrupted Vaginal Probiotic use
  Interventions: Drug: Vaginal Clindamycin Cream; Drug: Vaginal Probiotic

INTERVENTIONS:
Drug: Vaginal Clindamycin Cream — Vaginal Clindamycin Cream
  Other Names: dalacin c cream
Drug: Vaginal Probiotic — Vaginal Probiotic
  Other Names: dicoflor vaginal capsules

SUMMARY:
Vaginal Clindamycin Cream Plus Vaginal probiotic for treatment of Bacterial Vaginosis

DETAILED DESCRIPTION:
Vaginal Clindamycin Cream was used initially for treatment of Bacterial Vaginosis followed by Vaginal probiotic either in cnotinous or interrupted manner, then assessment of the results of treatment at different time intervals was done.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years
* has recurrent Bacterial Vaginosis

Exclusion Criteria:

* pregnancy
* use of other antmicrobial
* not provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
initial cure rate | 2 months
  number of women completely cured

SECONDARY OUTCOMES:
recurrence rate | 4,6,8and12 months
  number of women had recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim A EL sharkwy, Principal Investigator — FACULTY OF MEDICINE ,ZAGAZIG UNIVERSITY
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided